CLINICAL TRIAL: NCT01907347
Title: PHASE ANGLE PROJECT
Brief Title: Prognosis Value of Bioimpedance Analysis (BIA) Phase Angle at Admission in Intensive Care Unit (ICU) Patients
Acronym: PAP
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Collaborators: University Hospital, Clermont-Ferrand (Other); Erasme University Hospital (Other); Federal University of Pelotas (Other); Clinical Hospital Centre Zagreb (Other); University Hospital, Rouen (Other); Rabin Medical Center (Other); Vilnius University (Other); Stanley Dudrick's Memorial Hospital (Other); Clinica USP Palmaplanas (Unknown)
Responsible Party: Principal Investigator, Prof. Claude Pichard, Professor, MD, PhD, Head, Clinical Nutrition, University Hospital, Geneva
Other Study IDs: CEREH-13-022
Record Dates: First submitted 2013-07-13; First posted 2013-07-24 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Intensive Care Unit Patients
Keywords: intensive care unit (ICU); body composition; phase angle; mortality; nosocomial infection; bioimpedance analysis; nutrition
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICU patients

SUMMARY:
Critically ill patients feature a loss of fat-free mass (FFM) up to 440 g/day, which is associated with increased morbidity and prolonged recovery. In several clinical conditions, FFM or phase angle (PhA)derived from BIA have been associated with clinical outcome. However, solid data to support this association in ICU patients are lacking. Only one retrospective study of 51 ICU patients with acute respiratory failure correlated loss of active cell mass with mortality. In a pilot study performed in 55 ICU patients, the investigators observed that five kHz BIA PhA was significantly related to SOFA (r=0.38, P=0.03). The relation between PhA and mortality remains to be determined in ICU patients.

Classic ICU validated severity scores (e.g. Acute Physiology and Chronic Health Evaluation (APACHE), Sequential Organ Failure Assessment (SOFA), Simplified Acute Physiology Score (SAPS)) and recent nutritional scores have been developed to foresee the clinical outcome of ICU patients. Most of these scores are time consuming and suffer some degree of discriminative power (i.e. APACHE II and SAPS II are not validated in cardiovascular surgery patients).

PhA is reflecting intracellular status: altered intracellular water (ICW) to extracellular water (ECW) distribution is suggested by low PhA. PhA measurement does not require anamnestic parameters, body weight, and lab tests. It could easily, accurately and repeatedly measured at bedside. PhA has been correlated with the disease prognosis in HIV infection, hemodialysis, peritoneal dialysis, chronic renal failure and liver cirrhosis patients. These studies suggest that PhA may be useful in determining increased risk of morbidity in the ICU.

Computerized tomography (CT) images targeted on the 3rd lumbar vertebrae (L3) could accurately measure FFM13 and predict survival in cancer patients. Body composition evaluation by CT presents great practical significance due to its routine ICU use in the initial diagnosis or follow-up. The usefulness of measuring FFM with L3-targeted CT has never been evaluated in ICU patients.

Therefore, the investigators aim to conduct an international multicentre prospective observational study in ICU patients to assess the prognosis value of BIA PhA at admission, and to compare the performances of BIA and L3-targeted CT for FFM measurement.

ELIGIBILITY:
Inclusion Criteria:

* equal or more than 18 years
* expected ICU length of stay of more than 48 hours
* no readmission within the 48 hours following ICU discharge
* no Implanted Cardiac Devices
* no pregnancy or lactation
* affiliated to health insurance regimen
* informed consent by patient or next of kin.

Exclusion Criteria:

* age below 18 years
* expected ICU length of stay <48 hours
* readmission within the 48 hours following ICU discharge
* Implanted Cardiac Devices
* pregnancy or lactation
* non affiliated to health insurance regimen
* no informed consent by patient or next of kin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in medical and surgical intensive care units.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2014-08-15 (Actual); Study Completion 2014-08-31 (Actual)

PRIMARY OUTCOMES:
Mortality | 28-day after intensive care unit admission
  To determine the impact of phase angle at ICU admission, and phase angle changes during ICU stay, on 28-day mortality

SECONDARY OUTCOMES:
number of nosocomial infections | 28 day after the intensive care unit admission
  To determine the impact of phase angle at ICU admission, and phase angle changes during ICU stay, on the number of nosocomial infections 28 day after the intensive care unit admission.
length of mechanical ventilation | day 1 to day 28 after ICU admission
  To determine the impact of phase angle, and phase angle changes during ICU stay, at ICU admission on length of mechanical ventilation.
ICU length of stay | day 1 to ICU discharge or death
  To determine the impact of phase angle at ICU admission, and phase angle changes during ICU stay, on ICU length of stay.
hospital length of stay | day 1 to hospital discharge
  To determine the impact of phase angle at ICU admission, and phase angle changes during ICU stay, on hospital length of stay.
fat-free mass measurement by bioimpedance analysis and third lumbar vertebra-targeted computerized tomography | day 1 to day 28
  To compare bioimpedance analysis and third lumbar vertebra-targeted computerized tomography (CT) performances for fat-free mass measurement in the subgroup of patients being performed a routine abdominal CT.
ICU severity scores, APACHE II and SAPS II | within the 48 first hours of ICU stay
  Determine the relation between phase angle mortality predicted by the ICU severity scores, APACHE II and SAPS II

CONTACTS AND LOCATIONS:
Locations (10):
- Erasme University Hospital, Brussels, Belgium
- Universidade Federal de Pelotas, Pelotas, Brazil
- Univ. Hospital Center Zagreb, Zagreb, Croatia
- France (2):
  - Clermont-Ferrand University Hospital, Clermont-Ferrand
  - Rouen University Hospital, Rouen
- Rabin Medical Center, Petah Tikva, Israel
- Vilnius University Hospital, Vilnius, Lithuania
- Stanley Dudrick's Memorial Hospital, Skawina, Poland
- Clinica USP Palmaplanas, Palma de Mallorca, Spain
- Geneva University Hospital, Geneva, Switzerland

REFERENCES:
- [Derived] Thibault R, Makhlouf AM, Mulliez A, Cristina Gonzalez M, Kekstas G, Kozjek NR, Preiser JC, Rozalen IC, Dadet S, Krznaric Z, Kupczyk K, Tamion F, Cano N, Pichard C; Phase Angle Project Investigators. Fat-free mass at admission predicts 28-day mortality in intensive care unit patients: the international prospective observational study Phase Angle Project. Intensive Care Med. 2016 Sep;42(9):1445-53. doi: 10.1007/s00134-016-4468-3. Epub 2016 Aug 11. PMID 27515162